CLINICAL TRIAL: NCT05906888
Title: Invasive Mechanical Ventilation With Tracheostomy - an Observational Study on Patient-centered Outcomes
Brief Title: Weaning With Tracheostomy - an Observational Study on Patient-centered Outcomes
Acronym: Wean-Trach
Status: Completed | Type: Observational
Sponsor: Henrik Endeman (Other)
Collaborators: Franciscus &Vlietland (Other)
Responsible Party: Sponsor-Investigator, Henrik Endeman, Sponsor, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: W23.001
Record Dates: First submitted 2023-05-10; First posted 2023-06-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2024-11

CONDITIONS: Weaning Failure; Mechanical Ventilation; Patient-centered Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: It is largely undocumented how long it takes to wean from invasive mechanical ventilation (IMV) with tracheostomy and to what extend these patients suffer from dyspnea or discomfort and how often sputum retention occurs requiring burdensome endotracheal suctioning. In patients undergoing invasive mechanical ventilation via endotracheal tube, dyspnea is prevalent and associated with poorer quality of life and more symptoms of post-traumatic stress disorder (PTSD)

Objectives: The present study aims to assess the duration of the weaning period, and the prevalence and severity of dyspnea and discomfort in patients with tracheostomy-facilitated weaning.

Study design: Prospective observational multicenter cohort study. Study population: Tracheostomized critically ill patients weaning from IMV.

Main study parameters/endpoints:

Prevalence and severity of dyspnea and discomfort during weaning, duration of weaning with tracheostomy, frequency of endotracheal suctioning, time with tracheostomy, clinical outcomes, and mortality rates. Long term outcomes are the prevalence quality of life, PTSD, anxiety and fear.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Scheduled to start weaning from iMV, as per clinical decision

Exclusion Criteria:

* Deafness or Blindness
* Inability to speak or comprehend Dutch and English language
* Neuromuscular Disease
* Chronic positive pressure respiratory support at home (excluding night-time CPAP for sleep apnea)
* Support by Ventricular Assist Device or Extracorporeal life support (ECMO or ECCO2R) during tracheostomy-facilitated weaning phase.
* Tracheostomy primarily indicated for chronic upper airway obstruction or to secure airway patency due to persistent stupor/coma or swallowing disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a tracheostomy invasively ventilated in the ICUs of one of the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Daily dyspnea score during weaning | During repeated disconnection sessions in the first 28 days after initiation of weaning with tracheostomy, once daily an assessment is made using Visual Analog Scale for Dyspnea. (0-10). Higher scores indicate higher levels of dyspnea.
  The severity of dyspnea during disconnection from mechanical ventilation
Daily presence of dyspnea during weaning | During repeated disconnection sessions in the first 28 days after initiation of weaning with tracheostomy, once daily an assessment is made by asking communicative patients if they experience dyspnea.
  The severity of dyspnea during disconnection from mechanical ventilation; calculated as number of days with dyspnea, and percentage of weaning days with dyspnea.

SECONDARY OUTCOMES:
Weaning duration | From start weaning until separation attempt after tracheostomy placement until disconnection from the ventilator for ≥7 consecutive days, or ICU discharge, whichever comes first
  The time between the first disconnection session with tracheostomy and weaning
Mortality | From inclusion until 90 days after ICU discharge
  28-day, ICU- and in-hospital mortality
Health-related Quality of Life (HR-QoL) | 3 months after ICU discharge
  The HR-QoL, as measured with the EQ5D-5L questionnaire. High scores indicate a high level of perceived problems.
Health-related Quality of Life (HR-QoL) | 3 months after ICU discharge
  The HR-QoL, as measured with the EQ-VAS (0-100). High scores indicate a high level of self-reported HR-QoL.
Post-traumatic stress Disorder (PTSD) | 3 months after ICU discharge
  The presence PTSD-related symptoms, as measured with the IES-6 questionnaire
Anxiety and Depression | 3 months after ICU discharge
  The presence of long-term symptoms of anxiety and/or depression as measured with the Hospital-related Anxiety and Depression Scale (HADS) questionnaire.
Endotracheal suctioning | In the first 28 days after weaning initiation
  Number of endotracheal suctioning manoeuvres during the weaning phase
Daily discomfort score during disconnection session | During repeated disconnection sessions in the first 28 days after initiation of weaning with tracheostomy, once daily an assessment is made using Visual Analog Scale for Discomfort (0-10). Higher scores indicate higher levels of discomfort.
  The severity of discomfort
Duration of tracheostomy in situ | Within 90 days after tracheostomy placement

CONTACTS AND LOCATIONS:
Overall Officials: Evert-Jan Wils, MD PhD, Principal Investigator — Franciscus Gasthuis & Vlietland; Henrik Endeman, MD PhD, Study Director — Erasmus Medical Center
Locations (13):
- Netherlands (13):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia Ziekenhuis, Breda
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - St Anna ziekenhuis, Geldrop
  - Spaarne Gasthuis, Haarlem
  - Erasmus MC, Rotterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Haags Medisch Centrum Westeinde, The Hague
  - Elizabeth-Tweesteden Ziekenhuis, Tilburg

IPD SHARING:
Plan to Share IPD: Undecided